CLINICAL TRIAL: NCT05782374
Title: Studio Osservazionale Retrospettivo Multicentrico Sull'Utilizzo di Ibrutinib in Monoterapia o in Associazione a Immunochemioterapia Secondo Schema R-CHOP in Pazienti Adulti Con Diagnosi di PCNSL Ricaduto o Refrattario
Brief Title: Real World Data on Ibrutinib Use in PCNSL Rel/Ref
Acronym: ReWIPretro
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrés José Maria Ferreri, LYMPHOMA UNIT DIRECTOR, IRCCS San Raffaele
Other Study IDs: OSR REWIP
Record Dates: First submitted 2022-08-24; First posted 2023-03-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: PCNSL
Keywords: PCNSL; R-CHOP
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with r/r PCNSL: Adult patients diagnosed with relapsed or refractory PCNSL who in the period between August 2020 and May 2022 were candidates for treatment with ibrutinib alone or in combination with R-CHOP or R-CHOP like (in compassionate use, or off- label).
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — ibrutinib alone or in combination with R-CHOP or R-CHOP like

SUMMARY:
PCNSL is a rare and aggressive subtype of B lymphoma that has been recognized as a distinct disease entity in the latest edition of the WHO Classification of Tumors of Haematopoietic and Lymphoid Tissue and is defined as DLBCL that develops exclusively in the brain parenchyma, spinal cord, leptomeninges and eye. In patients under 70 years of age without severe comorbidities, first-line treatment with induction chemo-immunotherapy according to the MATRix scheme (Methotrexate, Cytarabine, Tiothepa, Rituximab) and subsequent consolidation with HDCT followed by ASCT achieved the best results in terms of PFS and OS. Data on patients enrolled in a randomized phase 2 study showed an OS of 70% at a median FU of 88 months. In patients> 70 years of age or with low KPS, the prognosis remains significantly lower in the younger population. Several population studies have shown a stable increase over the past 30 years in terms of PFS and OS in patients aged under 70 years, while in patients over 70 years or with KPS <70%, the survival curves are not satisfactory. in part because these patients are often referred to BSC alone, despite the benefit in PFS and OS demonstrated with HD-MTX-based treatments (≥1 g / m2) combined with oral alkylating agents or cytarabine in high doses.

DETAILED DESCRIPTION:
Historically, HDCT followed by ASCT has not been considered a feasible option for elderly patients, although recent data collected in the "real life" setting and a pilot study conducted in Germany demonstrate that maintenance of the dose intensity of HD-MTX and treatment completion with HDCT / ASCT-based consolidation are similar to those in clinical studies. However, 20 to 50% of newly diagnosed PCNSL patients do not achieve a complete response with currently available treatment regimens, highlighting the need for improved induction strategies. Furthermore, even after a complete response, patients with PCNSL may experience relapse, especially in the elderly. First-line treatment failure usually occurs (70-75% of cases) within the first two years and the prognosis of this population is extremely poor as demonstrated in a retrospective study of more than 250 patients with PCNSL R / R who reported median PFS and OS at first relapse / progression of 2.2 and 3.5 months, respectively. Similar results have also been highlighted in several prospective studies in which the PFS and OS curves are equivalent. There is currently no standard of treatment for the treatment of patients with PCNSL R/R. Data extrapolated from the long-term FU of a randomized phase 2 trial suggests that patients with relapses more than 36 months after the end of first-line methotrexate-based immuno-chemotherapy could benefit from a rechallenge with the same treatment. On the other hand, for patients refractory or with relapses within 36 months or not eligible for HD-MTX, the best therapeutic choice is represented by enrollment in a clinical trial. In the absence of this option, the therapeutic choice is based on the experience of phase 2 studies.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of DLBCL
* Disease localized exclusively in the CNS (brain, meninges, cranial nerves, eyes and / or spinal cord) both at first diagnosis and at failure
* Progressive or recurrent disease
* Previous treatment with high-dose methotrexate-based chemotherapy ± WBRT
* Age 18 - 80 years
* ECOG performance status 0-3
* Adequate hematopoiesis (platelets> 25,000 / mm3, hemoglobin> 8 g / dL, ANC> 1,000 / mm3), renal (serum creatinine <2 times UNL and creatinine clearance ≥40 mL / min), cardiac (VEF ≥50% ) and liver function (SGOT / SGPT <3 times UNL, bilirubin and alkaline phosphatase <2 times UNL).
* Patients who have been given treatment with ibrutinib, alone or in combination with immunochemotherapy, and who have or have not received the same.

Exclusion Criteria:

* Patients with concomitant extra-CNS disease at presentation or relapse
* Symptomatic coronary heart disease, cardiac arrhythmias not well controlled with drugs, or myocardial infarction within the past 6 months (New York Heart Association class III or IV heart disease)
* Any other serious medical condition that could compromise the patient's ability to adhere to treatment.
* Presence of any psychological, family, sociological or geographical condition that may hinder compliance with the study protocol and the follow-up program.
* In therapy with strong CYP3A inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with relapsed or refractory PCNSL who in the period between August 2020 and May 2022 were candidates for treatment with ibrutinib alone or in combination with R-CHOP or R-CHOP like (in compassionate use, or off- label).
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy in terms of overall rate of responses in patients treatment | 6MONTH
  To evaluate the efficacy in terms of overall rate of responses to treatment (ORR = sum of complete responses [CR] + partial responses [PR]) according to the IPCG 2005 criteria in a retrospective cohort of patients with relapsed / refractory PCNSL undergoing treatment with ibrutinib given as monotherapy or in combination with R-CHOP immuno-chemotherapy.

SECONDARY OUTCOMES:
Evaluate the effectiveness in terms of overall survival (OS); | 6MONTH
  Evaluate the overall survival (OS) after the treatment
Evaluate the effectiveness in terms of progression-free survival (PFS); | 6MONTH
  Verify the no progression of the lymphoma after the treatment
Verification of the safety of the ibrutinib monotherapy and in combination with R-CHOP | 6MONTH
  To evaluate the safety of ibrutinib administered alone and in combination with R-CHOP in the PCNSL R / R patient population;
To evaluate the role of consolidation therapy with high-dose chemotherapy | 6MONTH
  To evaluate the role of consolidation therapy with high-dose chemotherapy and autologous transplant or radiotherapy (ASCT or RT) and of ibrutinib maintenance therapy;
Frequency of invasive fungal infections after prophylactic antifungal therapy | 6MONTH
  Assess the frequency of invasive fungal infections and the effectiveness of prophylactic antifungal therapy in the patients treated with R-CHOP

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Louis DN, Perry A, Wesseling P, Brat DJ, Cree IA, Figarella-Branger D, Hawkins C, Ng HK, Pfister SM, Reifenberger G, Soffietti R, von Deimling A, Ellison DW. The 2021 WHO Classification of Tumors of the Central Nervous System: a summary. Neuro Oncol. 2021 Aug 2;23(8):1231-1251. doi: 10.1093/neuonc/noab106. PMID 34185076
- [Background] Ferreri AJM, Cwynarski K, Pulczynski E, Fox CP, Schorb E, Celico C, Falautano M, Nonis A, La Rosee P, Binder M, Fabbri A, Ilariucci F, Krampera M, Roth A, Hemmaway C, Johnson PW, Linton KM, Pukrop T, Gorlov JS, Balzarotti M, Hess G, Keller U, Stilgenbauer S, Panse J, Tucci A, Orsucci L, Pisani F, Zanni M, Krause SW, Schmoll HJ, Hertenstein B, Rummel M, Smith J, Thurner L, Cabras G, Pennese E, Ponzoni M, Deckert M, Politi LS, Finke J, Ferranti A, Cozens K, Burger E, Ielmini N, Cavalli F, Zucca E, Illerhaus G; IELSG32 study investigators. Long-term efficacy, safety and neurotolerability of MATRix regimen followed by autologous transplant in primary CNS lymphoma: 7-year results of the IELSG32 randomized trial. Leukemia. 2022 Jul;36(7):1870-1878. doi: 10.1038/s41375-022-01582-5. Epub 2022 May 13. PMID 35562406
- [Background] Schorb E, Fox CP, Kasenda B, Linton K, Martinez-Calle N, Calimeri T, Ninkovic S, Eyre TA, Cummin T, Smith J, Yallop D, De Marco B, Krampera M, Trefz S, Orsucci L, Fabbri A, Illerhaus G, Cwynarski K, Ferreri AJM. Induction therapy with the MATRix regimen in patients with newly diagnosed primary diffuse large B-cell lymphoma of the central nervous system - an international study of feasibility and efficacy in routine clinical practice. Br J Haematol. 2020 Jun;189(5):879-887. doi: 10.1111/bjh.16451. Epub 2020 Jan 29. PMID 31997308
- [Background] Kaji FA, Martinez-Calle N, Bishton MJ, Figueroa R, Adlington J, O'Donoghue M, Smith S, Byrne P, Paine S, Sovani V, Auer D, James E, Bessell EM, Grainge MJ, Fox CP. Improved survival outcomes despite older age at diagnosis: an era-by-era analysis of patients with primary central nervous system lymphoma treated at a single referral centre in the United Kingdom. Br J Haematol. 2021 Nov;195(4):561-570. doi: 10.1111/bjh.17747. Epub 2021 Aug 8. PMID 34368948
- [Background] Sieg N, Naendrup JH, Godel P, Balke-Want H, Simon F, Deckert M, Gillessen S, Kreissl S, Brockelmann PJ, Borchmann P, von Tresckow B, Heger JM. Treatment patterns and disease course of previously untreated Primary Central Nervous System Lymphoma: Feasibility of MTX-based regimens in clinical routine. Eur J Haematol. 2021 Aug;107(2):202-210. doi: 10.1111/ejh.13639. Epub 2021 May 26. PMID 33960535